CLINICAL TRIAL: NCT06078293
Title: A Feasibility Study of Home-based Exercise for Older Veterans With Serious Mental Illness
Brief Title: Home-based Exercise for SMI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving position and ending funding award early
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E5010-W; RX005010 (Other Grant/Funding Number: VA RRD)
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Serious Mental Illness
Keywords: schizophrenia; schizoaffective disorder; bipolar disorder; exercise; physical function; home-based
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise (Experimental): All participants in this single-arm trial will be in the exercise arm and receive the home-based exercise program.
  Interventions: Behavioral: Home-based Exercise Program

INTERVENTIONS:
Behavioral: Home-based Exercise Program — 12-week home-based exercise program that involves individualized exercise prescription and motivational health coaching calls.

SUMMARY:
Older Veterans with serious mental illness (schizophrenia, schizoaffective disorder, bipolar disorder) have reduced physical function (endurance, strength, mobility) that leads to lower quality of life. Exercise interventions are effective at improving physical function and could have a tremendous impact on this population. Despite the established benefits of exercise, there has been little work focused on improving multiple aspects of physical function in older Veterans with serious mental illness. The purpose of this study is to examine the feasibility and acceptability of a home-based exercise program for older Veterans with serious mental illness.

DETAILED DESCRIPTION:
Older Veterans with serious mental illness (schizophrenia, schizoaffective disorder, bipolar disorder) have significantly compromised physical function that leads to heightened rates of falls, hospitalizations, nursing home admissions, as well as early mortality. In fact, this population's physical function is compromised across multiple domains including mobility, endurance, and strength. Exercise is effective for increasing all domains of physical function (i.e., mobility, endurance, strength) in older Veterans. But, environmental difficulties (e.g., lack of transportation), low motivation, and medical issues affecting older Veterans with serious mental illness contribute to low engagement rates and high dropout rates in facility-based exercise programs. Individualized home-based exercise programs, which are safe and effective for older Veterans with health challenges, could address the main barriers to exercise in older Veterans with serious mental illness by promoting greater accessibility and individual tailoring. The purpose of this study is to evaluate the feasibility and acceptability of a 12-week home-based exercise program for older Veterans with serious mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Veteran enrolled at Providence VAHCS
* age 50 or older
* chart diagnosis of SMI (i.e., schizophrenia, schizoaffective disorder, or bipolar disorder)
* clinically stable defined as no inpatient psychiatric admission in the prior three months and no changes in psychiatric treatment in prior month
* medically safe to participate in exercise defined by no inpatient medical admission in prior three months and sign-off by Veteran's medical provider

Exclusion Criteria:

* diagnosis of Alzheimer's or related dementia
* presence of any medical contraindication for exercise including unstable angina, active proliferative diabetic retinopathy, oxygen dependence, or frank incontinence
* already participating in regular exercise defined as at least 60 minutes/week every week for prior six months or currently enrolled in a VA exercise or health promotion program

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Feasibility/Acceptability as measured by eligibility rate | Through completion of study (an average of 2 years)
  Eligibility rate when screening participants (12% is benchmark)
Feasibility/Acceptability as measured by number of participants enrolled in the study | Through completion of study (an average of 2 years)
  Number of participants enrolled in the study (benchmark is n=30)
Feasibility/Acceptability as measured by exercise session adherence | End of intervention (12 weeks)
  Percentage of exercise sessions completed out of total number prescribed (60% is benchmark)
Feasibility/Acceptability as measured by coaching call adherence | End of intervention (12 weeks)
  Percentage of motivational health coaching calls completed out of total scheduled (60% is benchmark)
Feasibility/Acceptability as measured by orientation session fidelity | End of intervention (12 weeks)
  Percentage of administered orientation sessions with a fidelity rating of at least adequate (80% is benchmark)
Feasibility/Acceptability as measured by coaching call session fidelity | End of intervention (12 weeks)
  Percentage of administered coaching calls with a fidelity rating of at least adequate (80% is benchmark)
Feasibility/Acceptability as measured by Client Satisfaction Questionnaire Total Score | End of intervention (12 weeks)
  Total score on the Client Satisfaction Questionnaire (CSQ-8), which is an 8-item measure with each item scored from 1-4 with higher scores representing greater acceptability of the intervention and the range of total scores spanning 8-32 (24 is benchmark).
Feasibility/Acceptability as measured by retention | Through completion of study (an average of 2 years)
  Percentage of participants that completed the endpoint assessment (70% is benchmark)
Feasibility/Acceptability as measured by assessment duration | End of intervention (12 weeks)
  Length of the assessment battery in minutes (60 minutes is benchmark)

CONTACTS AND LOCATIONS:
Overall Officials: Julia W Browne, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No